CLINICAL TRIAL: NCT02215993
Title: Sampling P2Y12 Receptor Inhibition With Prasugrel and Ticagrelor in Patients Submitted to Thrombolysis After Loading Dose of Clopidogrel
Brief Title: Sampling P2Y12 Receptor Inhibition With Prasugrel and Ticagrelor in Patients Submitted to Thrombolysis
Acronym: SAMPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Leonardo de Freitas Campos Guimarães, PhD student, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 51476
Record Dates: First submitted 2014-06-03; First posted 2014-08-13 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Acute Coronary Syndrome; Platelet Function
Keywords: Ticagrelor; Prasugrel; VerifyNow; Acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel (Active Comparator): After 300mg or 600mg loading dose of clopidogrel, this medication will be replaced by 60 mg prasugrel followed by 10mg per day for 30 days.
  Interventions: Drug: Prasugrel
- Ticagrelor (Active Comparator): After 300mg or 600mg loading dose of clopidogrel, this medication will be replaced by 180 mg ticagrelor followed by 90mg twice a day for 30 days.
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — After 8 to 6 hours after the dose of 300mg and 600mg respectively. Patients will be randomized in a 1:1 ratio to receive ticagrelor the dose of 180mg and maintained dose of 90 mg twice a day for thirty days or prasugrel dose of 60mg and maintained for thirty days at a daily dose of 10mg.
  Arms: Prasugrel
Drug: Ticagrelor — After 8 to 6 hours after the dose of 300mg and 600mg respectively. Patients will be randomized in a 1:1 ratio to receive ticagrelor the dose of 180mg and maintained dose of 90 mg twice a day for thirty days or prasugrel dose of 60mg and maintained for thirty days at a daily dose of 10mg.
  Arms: Ticagrelor

SUMMARY:
Introduction:

Platelet aggregation plays an important role in ischemic complications in patients undergoing to percutaneous coronary intervention (PCI). The addition of clopidogrel, as a second antiplatelet agent, to acetylsalicylic acid (ASA) was effective in reducing major cardiovascular events in patients with acute coronary syndrome (ACS).

However, approximately 30% of ACS patients are resistant to clopidogrel, representing a population of medically vulnerable and high risk for major cardiovascular events, including myocardial infarction (MI), stent thrombosis and death.

In the randomized trial TRITON, prasugrel compared to clopidogrel was more effective in significantly reducing the rates of MI (7.4% vs. 9.4%) and stent thrombosis (2.4% vs .1,1%) in patients with ACS, however, patients treated with prasugrel showed higher rates of bleeding (2.4 vs. 1.8%) and no difference in mortality. Upon analysis of subgroups is not recommended its use in patients with a history of stroke in those older than 75 years and weighing less than 60 kg.

The latest class of inhibitors of the P2Y12 receptor is the cyclopentyl-triazolopyrimidines represented by ticagrelor. Unlike the thienopyridines, ticagrelor interacts with the platelet receptors in a reversible way and has a beginning and peak of action faster.

The efficacy and safety of ticagrelor were evaluated in the study PLATO, where 18.624 patients with ACS were randomized to receive clopidogrel (75mg/day, with a loading dose of 300 to 600mg) or ticagrelor (90mg 2x/day with a loading dose of 180mg) The primary combined endpoint (mortality from vascular causes, MI or stroke) at 12 months was significantly lower in the ticagrelor (9.8% vs. 11.7%). There was no significant difference in the rates of major bleeding in both groups. Moreover, the isolated analysis of the rates of MI, vascular mortality and mortality from all causes showed statistically significant reduction in the ticagrelor users. In this study, the main adverse effects were dyspnea and bradycardia.

The assessment of platelet reactivity may allow the individualization of antiplatelet therapy. However, simply increasing the dose of clopidogrel in patients who persisted with high platelet reactivity was not able to reduce the combined endpoint of cardiovascular death, nonfatal myocardial infarction and stent thrombosis in six months.

In a population of patients with stable coronary artery disease, the substitution of clopidogrel for ticagrelor showed a rapid and persistent decrease in platelet aggregation measured by different laboratory methods. However, in patients with ACS subjected to PCI, the assessment of platelet aggregation after the replacement of clopidogrel for prasugrel or ticagrelor still requires evidence.

Objectives:

To evaluate the platelet response to ticagrelor and prasugrel in ACS patients with ST-segment elevation submitted to thrombolysis.

To evaluate security in follow up of 30 days.

Methods:

The study will be a prospective, randomized, single-center (São Paulo Hospital - Federal University of São Paulo), single-blind. The investigators will select 50 patients admitted with ACS with ST-segment elevation submitted to thrombolysis and who underwent cardiac catheterization between 3 to 24 hours in the case of reperfusion or immediately for rescue angioplasty. Blood sample for analysis of platelet aggregation through the system VerifyNow ®, shall be obtained immediately after the procedure on patients on clopidogrel for at least seven days in maintenance dose of 75mg or after 8 to 6 hours after the dose of 300mg and 600mg respectively. Patients will be randomized in a 1:1 ratio to receive ticagrelor the dose of 180mg and maintained dose of 90 mg twice a day for thirty days or prasugrel dose of 60mg and maintained for thirty days at a daily dose of 10mg. A new blood sample and analysis of platelet aggregation will be repeated after 2, 6 and 24 hours. The demographic and clinical data of this population will be collected in specific form and stored in databases for later analysis

ELIGIBILITY:
Inclusion Criteria:

* less than 75 years
* sign the consent form
* Acute coronary syndrome with ST-segment elevation submitted to thrombolysis

Exclusion Criteria:

* use of IIbIIIa inhibitor
* less than 60 kg
* history of stroke
* Patients with sick sinus syndrome, atrioventricular block second or third degree, not protected by pacemaker
* Chronic obstructive pulmonary disease
* Asthma
* Heart failure class III / IV
* renal replacement therapy
* Use of inducers (carbamazepine, phenytoin, phenobarbital, rifampicin and dexamethasone) or inhibitors (ketoconazole, itraconazole, ritonavir, saquinavir, clarithromycin) potent enzyme PYP3A

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Assessment of change in platelet aggregation | time 0, 2, 6 and 24 hours

SECONDARY OUTCOMES:
The number of incidence of bleeding | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Guimaraes, Principal Investigator — Federal University of São Paulo; Adriano Caixeta, Study Director — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, Brazil